CLINICAL TRIAL: NCT07109518
Title: Universal CD7 CART (uCD7 CART) Cell Injection in the Treatment of Relapsed or Refractory CD7 Positive Hematologic Malignancies: a Prospective, Single-arm, Single-center Clinical Study.
Brief Title: uCD7 CART for Relapsed or Refractory CD7 Positive Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025073
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia (AML); T Lymphoblastic Leukemia/Lymphoma
Keywords: Universal CD7 CAR-T (uCD7 CAR-T); Acute myeloid leukemia (AML); T lymphoblastic leukemia/lymphoma (T-ALL/LBL); Prospective study; Single-arm Clinical Study
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- uCD7 CART (Experimental): Two cohorts were established: (1) relapsed and refractory acute myeloid leukemia (AML) cohort; and (2) relapsed and refractory T lymphoblastic leukemia/lymphoma (T-ALL/LBL) cohort. A 3+3 dose escalation and rapid titration design was used to explore the maximum tolerated dose (MTD) for each cohort. During the accelerated titration phase, dose-limiting toxicity (DLT) assessments were performed for 1 subject per enrollment and dose escalation was performed until the first DLT event was observed. 3+3 dose escalation CAR-T dose groups were (1) 0.5×10^6 CART cells/kg; (2)1×10^6 CART cells/kg;(3) 3×10^6 CART cells/kg. DLT assessments will be performed first for the first 3 subjects at each dose level (including the last subject at the end of rapid titration) and then for 1 to 3 subjects per enrollment. Therefore, a minimum of 4 and a maximum of 12 patients are expected to be enrolled.
  Interventions: Biological: uCD7 CART

INTERVENTIONS:
Biological: uCD7 CART — Subjects screened to meet the requirements for uCD7 CART use will enter clinical trials. Subjects were assessed at baseline. Fludarabine (Flu) and cyclophosphamide (CTX) based preconditioning should be performed within 1 week prior to uCD7 CART infusion: Flu 30mg/m2 ×3 days; CTX 500mg/m2 ×3 days. The investigator can adjust the pretreatment regimen appropriately according to the condition of the subject, such as increasing the dose of CTX to 600mg/m2 ×3 days, increasing the application of cytarabine and etoposide. Infusion of uCD7 CART must be performed 24 hours after completion of chemotherapy preconditioning. uCD7 CART can be infused at D-1 if the requirement of 24 hours after completion of preconditioning is met.

SUMMARY:
The aim of this study was to evaluate the safety and efficacy of universal CD7 CART (uCD7 CART) cells in the treatment of patients with relapsed/refractory CD7-positive hematologic malignancies. In this single-arm, open-label, single-center, Phase 1 clinical trial, two cohorts were set up: (1) relapsed and refractory acute myeloid leukemia (AML) cohort; and (2) relapsed and refractory T lymphoblastic leukemia/lymphoma (T-ALL/LBL) cohort. Each cohort was planned to enroll 4-12 patients. uCD7 CART cells will be administered intravenously to explore the maximum tolerated dose (MTD) of each cohort using a 3+3 dose escalation and rapid titration design.

DETAILED DESCRIPTION:
This study will use universal CD7 CAR-T cells to treat CD7-positive relapsed or refractory hematological malignancies, especially AML and T-ALL/LBL patients. Two cohorts were established: (1) relapsed and refractory AML cohort; and (2) relapsed and refractory T-ALL/LBL cohort. A 3+3 dose escalation and rapid titration design was used to explore the MTD for each cohort. 3+3 dose escalation CAR-T dose groups were (1) 0.5×10^6 CART cells/kg; (2)1×10^6 CART cells/kg;(3) 3×10^6 CART cells/kg. A minimum of 4 and a maximum of 12 patients are expected to be enrolled. Fludarabine and cyclophosphamide-based preconditioning should be performed within 1 week prior to uCD7 CART infusion. uCD7 CART can be infused at D-1 if the requirement of 24 hours after completion of preconditioning is met. To evaluate the safety and efficacy of uCD7 CART cells in the treatment of patients with relapsed/refractory CD7-positive hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and <70 years, regardless of gender;
2. T-ALL/LBL was diagnosed according to the criteria of NCCN Clinical Practice Guidelines for Acute Lymphocytic Leukemia (2020.v1) and T-cell Lymphoma Clinical Practice Guidelines (2020.v1);
3. Patients diagnosed with AML with reference to the Guidelines for Diagnosis and Treatment of Adult Acute Myeloid Leukemia (2018 Edition) issued by the Health Commission;
4. Cytology confirmed that the tumor cells were CD7 positive.
5. Number of blasts in bone marrow ≥5% at screening (bone marrow morphology);
6. Complies with the diagnosis of relapsed/refractory AML, including any of the following conditions according to China Guidelines for Diagnosis and Treatment of Relapsed/Refractory Acute Myeloid Leukemia (2021 Edition):

   1. Primary refractory patients who did not achieve CR after two cycles of standard induction chemotherapy;
   2. CR after consolidation chemotherapy, relapse within 12 months;
   3. Relapse 12 months after remission but ineffective after conventional chemotherapy;
   4. 2 or more relapses;
   5. Relapse after hematopoietic stem cell transplantation.
7. Meet the diagnosis of relapsed/refractory T-ALL/LBL, including any of the following:

   1. Primary refractory patients who have not achieved complete response after two cycles of standard chemotherapy, or patients who have not achieved complete response after multi-line rescue chemotherapy;
   2. Relapse within <12 months after complete remission or ≥12 months after complete remission and fail to achieve complete remission induced by 1 or more cycles of standard treatment;
   3. Relapse after hematopoietic stem cell transplantation or relapse after CAR-T therapy at the same target;
8. Complies with diagnosis of other relapsed/refractory CD7 positive hematologic malignancies
9. Creatine clearance >60ml/min (Cockcroft and Gault formula); serum total bilirubin ≤3 times the upper limit of normal, serum ALT and AST ≤5 times the upper limit of normal range for patients without liver invasion;
10. Echocardiography showing left ventricular ejection fraction (LVEF) ≥50%;
11. Pulse oxygen saturation ≥92%;
12. The estimated survival time is more than 3 months;
13. ECOG score 0-2;
14. Subjects or their legal guardians voluntarily participate in this trial and sign the informed consent form.

Exclusion Criteria:

Subjects who met any of the following criteria were excluded from the study:

1. acute promyelocytic leukemia (APL);
2. Presence of a genetic syndrome such as Fanconi's anemia, Kostmann's syndrome, Shwachman syndrome or any other known syndrome of bone marrow failure;
3. Patients with uncontrolled active central nervous system leukemia (CNSL), i.e. cerebrospinal fluid grades CNS 2 and CNS 3;
4. Patients who have received anti-tumor therapy before infusion should be excluded if any of the following conditions are met:

   1. Systemic chemotherapy (except for pretreatment) within 1 week;
   2. For those who have received monoclonal antibody therapy, the last time of monoclonal antibody infusion is less than 5 half-lives or 4 weeks (whichever is shorter) at screening;
   3. Received donor lymphocyte infusion (DLI) within 6 weeks;
5. Presence of uncontrolled, serious, active infection at screening;
6. Patients with a history of serious heart disease, including: severe cardiac insufficiency (subjects with cardiac insufficiency of Class III or IV according to the New York Heart Association (NYHA) cardiac function classification standard), myocardial infarction within 12 months or cardiac angioplasty or stenting, unstable angina pectoris, ECG indicating significant QT interval prolongation (>480ms) or serious arrhythmia judged by the investigator;
7. Previous craniocerebral trauma, disturbance of consciousness, epilepsy, cerebral ischemia, cerebral vascular hemorrhagic disease and other medical history, and within six months of the need for drug treatment;
8. Patients with hepatitis B surface antigen (HBsAg) greater than 10E6 IU/mL, hepatitis C virus (HCV) antibody positive, human immunodeficiency virus (HIV) antibody positive, syphilis antibody test positive, EBER positive or EBV copy number greater than the upper limit of normal at screening;
9. Patients who must use steroid hormones during CAR-T infusion (except for local or inhaled steroid hormones); subjects who are receiving systemic steroid therapy before screening and need long-term systemic steroid therapy during treatment according to the investigator's judgment (except for inhaled or local use);
10. Subjects with autoimmune diseases requiring treatment, immunodeficient subjects, or subjects requiring immunosuppressive treatment;
11. Patients with acute graft-versus-host disease (GvHD) or moderate-to-severe chronic GvHD within 4 weeks prior to screening;
12. Patients with a history of allergy to any component of cell products;
13. Pregnant, lactating females, and subjects (male or female) of childbearing potential who are unable to use effective contraception within 1 year after cell infusion; male subjects who plan to become pregnant within 1 year after cell infusion; female subjects or partners who plan to become pregnant within 1 year after cell infusion;
14. Any condition that, in the opinion of the investigator, may increase the risk to the subject or interfere with the results of the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2028-06-28 (Estimated); Study Completion 2030-06-28 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） Any toxicity associated with uCD7 CAR-T cells, or life-threatening hematological or non-hematological toxicity. | 3 months after uCD7 CART cells infusion
  Any toxicity associated with uCD7 CART cells, or life-threatening hematological or non-hematological toxicity.
Number of adverse event of CD7 CART cells treatment | Participants will be followed for the duration of the treatment, an expected average of 24 months.

SECONDARY OUTCOMES:
Response rate in 3 months | 3 months after uCD7 CART cells infusion
Duration of remission (DOR） | Participants will be followed for the duration of the treatment, an expected average of 24 months.
  Time to first CR/CRi + PR (T-ALL/LBL) or CRc + PR (AML) to disease relapse or death due to leukemia after uCD7 CART infusion.
Event-free survival (EFS) | Participants will be followed for the duration of the treatment, an expected average of 24 months.
Leukemia-free Survival (LFS） | Participants will be followed for the duration of the treatment, an expected average of 24 months.
  Time from first CR/CRi (ALL/LBL) or CRc (AML) to relapse or death.
Proportion of patients receiving hematopoietic stem cell | Participants will be followed for the duration of the treatment, an expected average of 24 months.
Overall survival (OS) | Participants will be followed for the duration of the treatment, an expected average of 24 months.
  Time from the first infusion of uCD7 CART cells to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China